CLINICAL TRIAL: NCT01466504
Title: A Study of the Effect of Sorafenib or Regorafenib on p63 Expression and Keratinocyte Differentiation in Human Skin
Brief Title: Effect of Sorafenib or Regorafenib on P63 Expression and Keratinocyte Differentiation in Human Skin
Status: Terminated | Type: Observational
Why Stopped: Accrual did not meet expectations. Over nearly 2 years just 4 subjects were treated on study. The goal of 30 subjects was not attainable.
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: D11004
Record Dates: First submitted 2011-10-31; First posted 2011-11-08 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-03

CONDITIONS: Renal Cell Carcinoma; Hepatocellular Carcinoma; Colorectal Carcinoma
Keywords: P63; Sorafenib; Regorafenib; rash; skin toxicity; RCC; HCC; colorectal carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma, Hepatocellular; Colorectal Neoplasms; Ectrodactyly, Ectodermal Dysplasia, and Cleft Lip-Palate Syndrome 3; Exanthema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — skin biopsies will be performed using a 4mm biopsy punch. Participants will undero 2 skin biopsies - one prior to starting sorafenib or regorafenib, the other once rash develops. If a rash does not develop within 84 days a biopsy of normal skin will be done.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: skin punch biopsy — Skin biopsy prior to sorafenib or regorafenib treatment and when rash appears or 12 weeks into treatment.

SUMMARY:
Skin toxicity is a frequently observed side effect in the era of "molecularly targeted therapies". Skin toxicity following administration of protein kinase inhibitors such as sorafenib, regorafenib, lapatinib, sunitinib, and others can be debilitating to the patient, resulting in dose reduction and discontinuation of treatment. The mechanisms of skin toxicity induced by targeted chemotherapy, such as sorafenib or regorafenib, are poorly understood. Further research is warranted to better understand the pathophysiology of drug-related skin toxicity in this setting and develop correction strategies. This study tests the hypothesis that sorafenib and regorafenib interfere with p63 expression and keratinocyte differentiation and skin remodeling.

Eligible study participants will be evaluated clinically for evidence of skin toxicity during their visits to the outpatient Oncology clinics. Study participants will undergo skin biopsies before sorafenib or regorafenib treatment is initiated and once rash develops or 12 weeks into treatment with sorafenib or regorafenib. Skin biopsies will be performed in Oncology clinics by the study investigators and clinic support staff.

Study participants will undergo both skin biopsies regardless of whether they develop a rash. In patients who develop a rash the most representative lesion will be biopsied. A normal appearing area of skin will be biopsied in participants who do not develop a rash.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years old or older.
2. Histologically or cytologically confirmed diagnosis of a solid tumor (RCC, HCC, or colorectal cancer).
3. Participants are planning to initiate treatment with either sorafenib or regorafenib as a single chemotherapeutic agent
4. Able to swallow and retain oral medication and does not have any clinically relevant, active gastrointestinal disease or other condition that may significantly alter absorption, distribution, metabolism, or excretion of drugs.
5. Be able to provide written informed consent.

Exclusion Criteria

1. Patients who are or will be receiving other chemotherapeutic or molecularly targeted agents in addition to sorafenib or regorafenib
2. Concurrent moderate or severe chronic inflammatory skin condition (eczema, psoriasis)
3. Concurrent blistering skin disorder of any severity (such as pemphigus, bullous pemphigoid)
4. Connective tissue disorders with skin involvement (systemic lupus erythematosus, scleroderma, dermatomyositis, etc.)
5. Patients manifesting an allergic skin reaction (such as urticaria) or skin reaction as a complication of prior chemotherapy
6. Patients with skin lesions of infectious or non-infectious cause, precluding skin biopsy
7. Patients not willing to undergo skin biopsy
8. Patients who are pregnant or planning to become pregnant during their participation in the study.
9. Chemotherapy, targeted therapy, or biological therapy within two weeks of start of treatment.
10. Ability to give informed consent is compromised by cognitive and/or decisional impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer diagnosis of Renal Cell Carcinoma (RCC) or Hepatocellular Carcinoma (HCC) or Colorectal Carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2011-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
p63 expression levels | Week 12
  Tissue collection is done within 7 days prior to treatment and when rash develops. If no rash develops, normal skin will be biopsied at week twelve of treatment.

SECONDARY OUTCOMES:
Tumor response | Week 12
  Sorafenib and regorafenib potentially interfere with p63 expression and keratinocyte differentiation and skin remodeling. The extent of interference may indicate extent of tumor response.

CONTACTS AND LOCATIONS:
Overall Officials: Alexey V Danilov, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (2):
- United States (2):
  - Dartmouth-Hitchcock Medical Center, Norris Cotton Cancer Center, Lebanon, New Hampshire
  - White River Junction VA Medical Center, White River Junction, Vermont